CLINICAL TRIAL: NCT05874752
Title: Myocardial Function Assessment in Patients With Coronary Artery Disease Using Noninvasive Myocardial Work
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-029-01
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Noninvasive Myocardial Work; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nonsignificant coronary artery stenosis group: Exclusion criteria: ≥70% proximal luminal stenosis in at least one major coronary vessel based on coronary angiography
  Interventions: Diagnostic Test: Transthoracic echocardiography
- significant coronary artery stenosis group: Defined as ≥70% proximal luminal stenosis in at least one major coronary vessel based on coronary angiography
  Interventions: Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — noninvasive myocardial work

SUMMARY:
Noninvasive pressure-strain loop (PSL) derived myocardial work (MW) are more sensitive than conventional echocardiographic parameters in quantitative assessment of early myocardial dysfunction. The aim of this study was to assess left ventricular (LV) myocardial function in symptomatic patients with coronary artery disease using the promising method.

Methods: Transthoracic echocardiography was performed on patients with angina or equivalent symptoms before coronary angiography. Images were stored and imported into the software for further offline analysis of PSL-based MW. MW analysis were carried out on each patient for global and regional myocardial function assessment.

ELIGIBILITY:
Inclusion Criteria: Patients who were hospitalized for coronary angiography with angina or equivalent symptoms.

-

Exclusion Criteria: Acute coronary syndrome, left main stem coronary disease, left ventricular ejection fraction (LVEF) below 55%, observed resting regional wall motion abnormalities (RWMAs), non-sinus rhythm, intraventricular block, previous cardiac surgery, severe valvular heart disease, hypertrophic cardiomyopathy, myocarditis, pericardial diseases, pulmonary hypertension, and poor image quality.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were hospitalized for coronary angiography with angina or equivalent symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
myocardial function | baseline (before coronary angiography)
  noninvasive myocardial work indices

CONTACTS AND LOCATIONS:
Overall Officials: Yingmei Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No